CLINICAL TRIAL: NCT07006467
Title: Study to Evaluate the Feasibility of the Resorbable Fibrillated Scaffold (RFS) in Arterial Lesions Below the Knee, in Patients With Critical Limb Ischemia
Brief Title: Initial Feasibility Study of the STENTiT Resorbable Fibrillated Scaffold (RFS). The RFS is Intended to Restore Lumen Patency and Blood Flow to Infrapopliteal Arteries. The RFS is a Fully Electrospun Tubular Device With a Fibrillated Microarchitecture and Designed for Transcatheter Delivery
Acronym: VITAL-IT 1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stentit (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-10001 VITAL-IT 1
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Critical Limb Ischemia (CLI)
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RFS arm (Experimental): Peripheral transluminal angioplasty with the RFS of the below the knee vasculature
  Interventions: Device: Implantation of RFS

INTERVENTIONS:
Device: Implantation of RFS — Percutaneous transluminal implantation of the RFS in the infrapopliteal lesion

SUMMARY:
This is the First-In-Human feasibility study of the RFS for below the knee lesions in subjects who experience critical limb ischemia due to the peripheral artery disease. The aim of this study is to investigate if the RFS can be implanted safely and with technical success. Up to 10 subjects will be treated with the RFS at one investigational site. Lesions within the inflow trajectory or side branches may be treated with institutions standard of care prior to treatment of the target lesion. This may include usage of POBA, BMS, DCB, or DES. The target lesion will be predilated with POBA.

Device safety will be assessed throughout the clinical investigation, with primary safety endpoints defined as freedom from Major Adverse Limb Events (MALE) at 30 days follow-up. In addition, MALE at 3-, 6-, 12-, and 24- months follow-up, all adverse events, serious adverse events and all device deficiencies will be captured as secondary endpoints.

Device performance will be based on technical success of the implantation defined as successful delivery and deployment with a residual area stenosis of ≤50% as determined on final perioperative IVUS. Primary patency at day of discharge, 30-days, 3-, 6-, 12-, and 24- months follow up will be captured as secondary performance endpoint and are based on duplex ultrasound for all timepoints and angiography and IVUS at 6-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria:

  1. Subject must provide written informed consent prior to any clinical investigation related procedures.
  2. Subject is willing and able to comply with the study procedures, and follow-up schedule.
  3. Subject has Critical Limb Ischemia (CLI), Rutherford Becker Clinical Category 4 or 5
  4. Subject must be at least 18 years of age.

     Anatomical inclusion criteria:
  5. Target lesion located in the tibioperoneal trunk, or 2/3 proximal part of the anterior tibial artery, posterior tibial artery or peroneal artery.
  6. Only one target lesion per subject is included, other lesions can be treated per institution's standard of care.
  7. At least one infrapopliteal branch without an angiographic significant lesion (≥50% diameter stenosis by angiography).
  8. Vessel diameter of 3.0 mm to 3.4 mm. Quantitative imaging (IVUS and angiography) will be used to aid accurate sizing of the vessels.
  9. Target lesion length ≤ 18 mm.
  10. Target lesion of ≥70% diameter stenosis, per angiographic assessment at the time of the procedure.
  11. Target lesion is in an area that may be stented without blocking access to subject main branches, i.e ≥2 mm distanced from any bifurcation.
  12. Successful antegrade crossing of the target lesion

Exclusion Criteria:

* General exclusion criteria:

  1. Subject is currently participating in another clinical investigation that has not yet reached the primary endpoint.
  2. Pregnant or nursing subjects or with planned pregnancy during the clinical investigation follow-up period.
  3. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements.
  4. Incapacitated individuals, as defined as persons who are mentally ill, mentally handicapped, or individuals without legal authority, are excluded from the study population.
  5. Subject has known hypersensitivity or contraindication to device material and its degradants (poly (L-lactide), poly (glycolic acid), lactic acid, and glycolic acid) that cannot be adequately pre-medicated. Subject has known contrast sensitivity that cannot be adequately pre-medicated.
  6. Subject has known allergy hypersensitivity or contraindication to aspirin; or to ADP antagonists such clopidogrel, prasugrel or ticagrelor; or to anticoagulants such as heparin or bivalirudin, and therefore cannot be adequately treated with study medications.
  7. Subject with planned surgery or procedure necessitating discontinuation of antiplatelet medications, within 3 months after index procedure.
  8. Subject has life expectancy ≤ 1 year.
  9. Subject has had a stroke within the previous 3 months with residual Rankin score of ≥2.
  10. Subject has renal insufficiency as defined as an estimated GFR < 30ml/min per 1.73m2
  11. Subject has platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC < 3,000 cells/mm3, or hemoglobin < 9.0 g/dl.
  12. Subject has known serious immunosuppressive disease (e.g. human immunodeficiency virus), or has severe autoimmune disease, that requires chronic immunosuppressive therapy (e.g. systemic lupus erythematosus, etc.), or subject is receiving immunosuppression therapy for other conditions. Subjects treated for HIV (Human Immunodeficiency Virus) and who have undetectable viral load, such that their immune system is not considered compromised, are eligible.
  13. Subject has Body Mass Index (BMI) < 18.
  14. Subject has a known coagulation disorder with increased risk of arterial thrombosis. Subject with deep vein thrombosis and disorders that increase the risk of deep vein thrombosis can be included in the study.
  15. Subject who requires thrombolysis as a primary treatment modality or requires other treatment for acute limb ischemia of the target limb.
  16. Subject has previously had or requires surgical revascularization involving any vessel of the ipsilateral extremity.
  17. Subject has signs or symptoms of advanced limb infection or septicemia (fever > 38.5 degrees Celsius, WBC > 15,000 cells/microliter, hypotension) at the time of assessment.
  18. Subject with extensive tissue loss salvageable only with complex foot reconstruction or non-traditional transmetatarsal amputation.

      Anatomic exclusion criteria:
  19. Subject has tandem lesions at the target lesion site (plaque free zone < 2 cm)
  20. Pre-dilatation of the target lesion at the time of study intervention did not reach <50% residual diameter stenosis by angiography.
  21. Target lesion that has prior metallic stent implant.
  22. Failed PTA of target lesion ≤ 60 days prior to the procedure date.
  23. The target vessel has another significant lesion (≥50% diameter stenosis by angiography).
  24. Significant stenosis (≥50% stenosis) lesion in a distal outflow artery that would be perfused by the target vessel and that requires treatment at the time of the index procedure.
  25. Subject has angiographic evidence of, thrombus, thromboembolism or atheroembolism in the ipsilateral extremity.
  26. Unsuccessfully treated proximal inflow limiting arterial stenosis or inflow-limiting arterial lesions left untreated.
  27. Aneurysm in the iliac, common femoral, superficial femoral, popliteal or target artery of the ipsilateral extremity.
  28. Target lesion has a high probability that atherectomy will be required at the time of index procedure for treatment of the target vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety: Freedom from Major Adverse Limb Event (MALE) + Perioperative Death (POD) | 30 day follow-up
  Safety:
  Freedom from Major Adverse Limb Event (MALE) + Perioperative Death (POD)
  * MALE includes:
  * Above ankle amputation in index limb or Any target lesion re-intervention at 30-day follow-up
  * POD includes:
  Mortality at 30 days follow-up
Performance: Number of patients with Technical Success | perioperative
  Technical success is defined as successful delivery and deployment of the RFS to the target lesion resulting in a final residual area stenosis of ≤50% as assessed on intravascular ultrasound (IVUS).
  * Successful delivery is defined as reaching the target lesion and successful withdrawal of the delivery catheter.
  * Successful deployment is determined by the achieved pressure (in atm) on the balloon combined with visual assessment of the balloon inflation on angiography.
  * ≤50% residual area stenosis is verified by independent Core Lab analysis of perioperative IVUS measurements. If IVUS is not available or insufficient, ≤30% final residual diameter stenosis at perioperative angiography will be used to assess Technical Success.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Universiteit Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol